CLINICAL TRIAL: NCT00195481
Title: A Post Marketing Surveillance Looking at Safety of Rapamune (Sirolimus) in Indian Population Undergoing de Novo Renal Transplantation.
Brief Title: Study Evaluating Sirolimus in Kidney Transplant Recipients in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0468H-101543
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Kidney Failure; Graft vs Host Disease
Keywords: Kidney; Transplant
MeSH Terms: conditions — Renal Insufficiency; Graft vs Host Disease | interventions — Sirolimus

INTERVENTIONS:
Drug: Rapamune

SUMMARY:
To determine the safety of sirolimus tablets in renal allograft recipients in a postmarketing surveillance setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients in End Stage Renal Disease who are above 13 years of age and weigh more than 40 kilograms.
* Patients scheduled to receive a kidney from a cadaveric donor, from a living unrelated donor or from a living related donor.

Exclusion Criteria:

* Evidence of major infections at the time of sirolimus administration
* Use of any investigational drug or treatment up to 4 weeks prior to enrolling in the study and during the treatment phase.
* Females who are pregnant, breast feeding or in reproductive age group and not using a medically acceptable form of contraception

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- India (4):
  - Bangalore, Karnataka
  - Saket, South Delhi
  - Chennai, Tamil Nadu
  - New Delhi